CLINICAL TRIAL: NCT01125995
Title: A Randomized Phase III Trial for Timing of Radiation in Concurrent Chemoradiation for Limited Stage Small-cell Lung Cancer
Brief Title: Early Versus Late Concurrent Chemoradiation for Limited Stage Small-cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Keunchil Park, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-02-016
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Small Cell Lung Cancer
Keywords: limited disease
MeSH Terms: conditions — Small Cell Lung Carcinoma

ARMS (2):
- late CCRT (Active Comparator): radiotherapy start on day one of the third cycle of chemotherapy
  Interventions: Radiation: late CCRT
- Early CCRT (Experimental): Radiotherapy start on day 1 of 1st cycle of chemotherapy
  Interventions: Radiation: early CCRT

INTERVENTIONS:
Radiation: early CCRT — 1. patients will be received with 4 cycles of etoposide 100mg/m2 D1-3 & Cisplatin 70mg/m2 D1.
  2. radiotherapy start from day 1 of 1st chemotherapy cycle and complete 5250cGy/25fraction (daily one fraction, 210cGy).
  Arms: Early CCRT
Radiation: late CCRT — 1. patients will be received with 4 cycles of etoposide 100mg/m2 D1-3 & Cisplatin 70mg/m2 D1.
  2. radiotherapy start from day 1 of the third cycle of EP chemotherapy and complete 5250cGy/25fraction (daily one fraction, 210cGy).
  Arms: late CCRT

SUMMARY:
The purpose of the study is to evaluate the efficacy and toxicity of different timing of concurrent chemoradiation in the treatment of limited disease status Small-cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed small-cell lung cancer
* limited disease status
* with evaluable disease
* 18 years or older
* ECOG performance status 0,1,2
* expected survival time should be 12 weeks or longer
* Adequate organ function as evidenced by the following; Absolute neutrophil count > 1.5 x 109/L; platelets > 100 x 109/L; total bilirubin ≤1.5 UNL; AST and/or ALT < 5 UNL; creatinine clearance ≥ 50mL/min
* Written informed consent form

Exclusion Criteria:

1. Uncontrolled systemic illness such as DM, CHF, unstable angina, hypertension or arrhythmia
2. Patients with active infection requiring antibiotics
3. Pregnant or nursing women ( Women of reproductive potential have to agree to use an effective contraceptive method)
4. Prior history of malignancy within 5 years from study entry except for a adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer, well-treated thyroid cancer
5. previous history of chemotherapy or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2003-06; Primary Completion 2011-07 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
complete response rate | 6 months

SECONDARY OUTCOMES:
overall survival | 36 months
objective response rate | 6 months
Progression-free survival | 36 months
toxicity by NCI common toxicity version 2.0 | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Keunchil Park, Principal Investigator — Samsung Medical Center
Locations (2):
- South Korea (2):
  - Keunchil Park, Seoul
  - Asan Medican Center, Seoul